CLINICAL TRIAL: NCT03883230
Title: A Multi-centre, Controlled, Prospective Cohort Study Investigating the Accuracy of the Glycologic Limited Test Kit to Detect Bacterial Infection in Chronic and Delayed-healing Wounds.
Brief Title: Wound Infection Detection Evaluation, WIDE
Acronym: WIDE
Status: Completed | Type: Observational
Sponsor: Cumbria Partnership NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CP1713
Record Dates: First submitted 2019-02-15; First posted 2019-03-20 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Wound Infection Bacterial; Ulcer Foot; Diabetic Foot; Diagnostic Self Evaluation
MeSH Terms: conditions — Foot Ulcer; Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic wound: All patients will have a Glycologic infection detection test (GLYWD) taken. For this, a standard CE-marked sterile swab is used to take a wound exudate sample. This is then inserted in the GLYWD detection tube device. The device will contain two separate reagents, one in the clear plastic vial end and the other in the foil-sealed compartment. The sterile swab with the wound exudate sample will be pushed into the device, breaking the foil-sealed compartment and allowing the reagents to mix with the sample. the result of the test - to see if there is a bacterial infection present in the wound - is observed up to ten minutes later.
  Interventions: Diagnostic Test: GLYWD

INTERVENTIONS:
Diagnostic Test: GLYWD — As mentioned in the group description, GLYWD is a plastic test tube and a chromatic test that contains two solutions. When combined with a wound exudate and incubated at RT, it will change colour to red if there is a pathological bacterial wound infection present.

SUMMARY:
Chronic wounds, such as diabetic foot ulcers, place a huge burden on healthcare systems and can lead to complications with high morbidity, particularly if the wound if infected. In parallel, there is pressure to reduce the use of antibiotics in order to minimise the risk of antimicrobial resistance. The Glycologic wound detection kit (GLYWD) is a point-of-care test, designed to provide guidance to clinical staff as to whether a chronic wound is infected or not. In this prospective cohort study the premise of this mode-of-action is evaluated. GLYWD will be applied in conjunction with clinical opinion and microbiological testing to determine if there is concordance between the different diagnostic approaches, and if applicable how they may differ in certain patients' wounds.

DETAILED DESCRIPTION:
The occurrence of diabetic foot ulcer (DFU) is a common complication of diabetes with enormous cost implications, totalling £650 million per year once associated morbidity is taken into account (NHS Diabetes report). Bacterial infection of wounds carries the risk of further degenerative complications including cellulitis, necrotising fasciitis, and sepsis (Grothier, 2015). Specific wounds, such as diabetic foot ulcers may lead to amputation if osteomyelitis develops. An additional undesirable effect of infection of wounds is that it delays - or stops altogether - the wound healing process (Halbert et al, 1992).

Detection of DFU infection remains reliant on clinical judgement. For example, imaging modalities such as MRI do not perform better than clinical appraisal in terms of sensitivity and specificity when it comes to detecting osteomyelitis (Dinh et al, 2008). O'meara and colleagues (2006) concluded from a systematic review on clinical examination, sample acquisition and sample analysis in DFUs that there is a lack of evidence regarding what samples should be taken and how they should be analysed. They did suggest that semi-quantitative sample analysis - a category that the Glycologic detection kit (called GLYWD) would fall under - may be a useful alternative to quantitative analysis. Quantitative detection of infection is still undertaken by swabbing the wound and then culturing the pathogens in a microbiology laboratory. Obtaining these results generally takes days; even molecular profiling does not give an instant result. Microbiological counts and species identification do not necessarily reflect infection as defined by other assessments, as demonstrated by Gardner et al (2014).

Clinical guidelines stipulate that the only available laboratory-based diagnostic option, microbiological testing, should only be used to identify the pathogen strain in clinically confirmed infection. Therefore, clinical opinion is the mainstay of predicting and diagnosing infection (NICE, 2008, 2015). The lack of a simple cost-effective and repeatable testing method may have three consequences: 1) lack of uniformity in diagnosis, due to differences in clinical judgement, which in turn may result in 2) over-diagnosis of infection with inappropriate prescription of antibiotics or antimicrobial dressings, or 3) late presentation of patients with systemic signs and spreading cellulitis or osteomyelitis requiring hospital admission and treatment with intravenous antibiotics or emergency surgery.

The provision of a rapid, reliable, sensitive and relatively low cost infection detection test kit for infection, which can be used at point-of-care, has the potential to provide the NHS with significant cost savings as well as improving the outcomes for patients. Therefore, in this study the Glycologic diagnostic wound infection detection test (GLYWD) is evaluated against clinical opinion and microbiological diagnostics to determine if it is an effective tool for the rapid detection of chronic wound infection.

ELIGIBILITY:
Inclusion Criteria:

* - Adult patients aged > 18 years
* Patients with recurrent wounds, including multiple wounds, are eligible (including patients who have concluded participation in this study for one wound, but have another wound in another location).
* If infection occurs, and/or antibiotics applied, whilst in study then this is not deemed an exclusion criterion.
* DFU element: Clinical diagnosis of Diabetic Foot Ulcer (DFU) with wound duration > 30 days.
* Other Other chronic and delayed-healing wounds element: Clinical diagnosis of a chronic or delayed-healing wound, with the wound present for at least 6 weeks. To include:

  * Pressure ulcer
  * Leg ulcer (can be venous, mixed or arterial in nature)
  * Non-diabetic foot ulcer
  * Post-operative wound
  * Trauma or other non-surgical wounds

Exclusion Criteria:

* - Aged < 18 years
* Any reasons for the patient being unable to follow the protocol, including lack of mental capacity to consent to taking part in the study.
* The patient has concurrent (medical) conditions that in the opinion of the investigator may compromise patient safety or study objectives
* DFU element only:
* Confirmed and ongoing wound infection at baseline which is already being treated with systemic antibiotics.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic non-infected Diabetic Foot Ulcers (DFU) or other chronic and delayed-healing wounds will be recruited into the study. Patients will be recruited from the adult population seen routinely by the evaluation clinical staff.
Sampling Method: Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
GLYWD test result | 10 minutes
  Result of diagnostic testing of wound with GLYWD

SECONDARY OUTCOMES:
Microbiology result of wound swab | 2 days
  The wound will be assessed with standard microbiological techniques. After 2 days incubation at 37C and 5% CO2, the types of bacteria isolated and grown in the swab sample will be reported. This will be using standard Colony Forming Units (CFU)
Clinician's wound characterization | 1 minute
  A clinician's scoring of wound characteristics for infection (absent, possible infection, definite infection), and the three hallmark signs of infection, namely: erythema (-, +, ++) purulence (-, +, ++), odour (none, mild, moderate, severe)

CONTACTS AND LOCATIONS:
Overall Officials: Leon Jonker, PhD, Principal Investigator — Cumbria Partnership NHS Trust, UK
Locations (1):
- Research & Development Department, Carlisle, Cumbria, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not applicable. We'll share the anonymised raw data -with individual but not with personal identifiable data included- with the journal that we submit results to.